CLINICAL TRIAL: NCT01760122
Title: A Phase 3, Randomized, Multi-center, Active-controlled, Open-label Study to Evaluate the Efficacy and Safety of Peginterferon Alfa-2b (40kD, Y Shape) in Chinese Chronic Hepatitis B Patients.
Brief Title: Efficacy and Safety of Peginterferon Alfa-2b in HBeAg Positive Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB1211IFN
Record Dates: First submitted 2012-12-30; First posted 2013-01-03 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Hepatitis B
Keywords: peginterferon; HBeAg Positive; Chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ypeginterferon Alfa-2b (Experimental)
  Interventions: Drug: Ypeginterferon alfa-2b
- Pegasys (Active Comparator)
  Interventions: Drug: Pegasys

INTERVENTIONS:
Drug: Ypeginterferon alfa-2b — sc, qw, 48 weeks.
  Arms: Ypeginterferon Alfa-2b
Drug: Pegasys — sc, qw, 48 weeks.
  Arms: Pegasys

SUMMARY:
This study is aimed to assess the efficacy and safety of Peginterferon alfa-2b (40kD, Y-shape), in a dose of 180μg/week, in chronic hepatitis B patients, and collects sufficient evidences for the listed of the studied drug.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18~65 years.
* Serum HBsAg or HBV DNA positive for at least 6 months.
* Serum HBsAg and HBeAg are both positive, HBV DNA ≥ 20,000IU/ml at screening.
* 2×ULN≤ ALT ≤10×ULN at screening (ULN=upper limit of normal).
* Pregnancy tests of female patients must be negative. All patients with effective birth control measures during treatment period and 6 months after the treatment.

Exclusion Criteria:

* Pregnant or lactating women.
* Mental disorder or physical disability.
* Interferon treatment history or using nucleos(t)ide analogue for chronic hepatitis B treatment within the previous 6 months.
* ANC < 1500/mm3, or PLT < 90,000/mm3.
* Co-infection with HAV, HIV, HCV, HDV, or HEV.
* Both of HBsAg and anti-HBs are positive, or both of HBeAg and anti-HBe are positive at screening.
* Child-Pugh ≥ B, or other evidence of hepatitis decompensation (e.g.: prothrombin time prolonged more than 3 seconds, TBil > 2ULN, Alb<35g/L).
* Chronic hepatitis caused by any other reason except hepatitis B.
* Hepatocarcinoma or suffering from any other malignant tumor.
* Not well-controlled endocrine diseases (e.g.: thyroid dysfunction, diabetes mellitus)
* Significant function damage in any major organs (e.g.: heart, lung, kidney).
* Other Conditions which in the opinion of the investigator precluding enrollment into the study (e.g.: poor compliance).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2013-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBeAg seroconversion at week72 | 24 weeks after the cessation of treatment

SECONDARY OUTCOMES:
Proportion of Patients with HBeAg seroconversion at week 12,24,48 | week 12, 24, 48 from treatment starting
Proportion fo patients with HBeAg undetectable at week 12, 24, 48, and 72. | week 4, 12, 24, 48 and 72 from treatment starting
Average of HBV DNA decline level at week 12, 24,48 and 72 | week 12, 24, 48 and 72 from treatment starting
Average of HBsAg decline level at week 12, 24, 48 and 72, and Proportion of patients with HBsAg undetectable and HBsAg seroconversion at week 12, 24, 48 and 72. | week 12, 24, 48 and 72 from treatment starting
Proportion of patients with ALT normalization at week 12,24, 48 and 72. | week 12, 24, 48 and 72 from treatment starting

CONTACTS AND LOCATIONS:
Overall Officials: Wang Guiqiang, Ph.D, Principal Investigator — Peking University First Hospital
Locations (43):
- China (43):
  - Xiamen Hospital of T.C.M, Xiamen, Fujian
  - Beijing University Shenzhen Hospital, Shenzhen, Guangdong
  - 302 Military Hospital, Beijing
  - Beijing Ditan Hospital Capital Medical University, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Beijing Youyi Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - First Affiliated Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central-south University, Changsha
  - Xiangya Second Hospital, Central-south University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Southwest Hospital, Chongqing
  - Fuzhou Infectious Disease Hospital, Fuzhou
  - Guangzhou Eighth People's Hospital, Guangzhou
  - Nanfang Hospital, Guangzhou
  - First Affiliated Hospital of Guangxi Medical University, Guilin
  - First Affiliated Hospital, Zhejiang University, Hangzhou
  - Second Affiliated Hospital of Harbin Medical University, Harbin
  - Jinan Infectious Disease Hospital, Jinan
  - First Affiliated Hospital of Lanzhou University, Lanzhou
  - 81 Military Hospital, Nanchang
  - First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Second Hospital of Nanjing, Nanjing
  - 85 Military Hospital, Shanghai
  - Huashan Hospital, Shanghai
  - Ruijing Hospital, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Shenyang Sixed People's Hospital, Shenyang
  - Third Affiliated Hospital, Hebei Medical University, Shijiazhuang
  - First Affiliated Hospital, Shanxi University, Taiyuan
  - Tianjin Third Central Hospital, Tianjin
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - First Affiliated Hospital of Wenzhou Medical College, Wenzhou
  - Tongji Hospital, Huazhong University of Science & Technology, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tangdu Hospital, Fourth Military Medical University, Xi'an
  - Xijing Hospital, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Provincial People's Hospital, Zhengzhou